CLINICAL TRIAL: NCT01247337
Title: Intra-hepatic Chemotherapy With Oxaliplatin Every Second Week in Combination With Systemic Gemcitabine and Capecitabine in Combination With Cetuximab in Patient With Non-resectable Liver Metastases From Cholangiocarcinoma. A Phase II Trial.
Brief Title: Intra-hepatic Chemotherapy in Patient With Non-resectable Liver Metastases From Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dorte Nielsen (Other)
Responsible Party: Sponsor-Investigator, Dorte Nielsen, Responsible Party was entered in the old format as Dorte Nielsen, professor DMSci, Department of Oncology, Herlev Hospital., Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI 1003
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Oxaliplatin; Capecitabine; Gemcitabine; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm chemotherapy treatment (Experimental)
  Interventions: Drug: Oxaliplatin, capecitabine, gemcitabine, cetuximab; Drug: Oxaliplatin, capecitabine, gemcitabine cetuximab

INTERVENTIONS:
Drug: Oxaliplatin, capecitabine, gemcitabine, cetuximab — Intrahepatic oxaliplatin
Drug: Oxaliplatin, capecitabine, gemcitabine cetuximab — Oxaliplatin given intravenous

SUMMARY:
A phase II trial evaluating intra-hepatic chemotherapy with oxaliplatin every second week in combination with systemic gemcitabine and capecitabine in combination with cetuximab in patient with non-resectable liver metastases from cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:• Informed consent

* Age > 18 years
* Performance status 0-1; expected survival ≥ 3 months
* Patient with histologically or cytologically adenocarcinoma developed from cells in the gall bladder, extra- or intrahepatic bile ducts or malignant cells consistent with above mentioned and radiologic findings consistent with cholangiocarcinoma
* Liver metastases not suitable for surgery or other local treatment
* Extrahepatic disease should be excluded by PET-CT-scan.
* Prior treatment with chemotherapy or no progression on first line treatment
* Metastases < 70 % of the liver
* neutrophile granulocytes ≥ 1.5 x 109/l og thrombocytes ≥ 100 x 109/l
* bilirubin < 2.0 x UNL (upper normal limit).
* creatinine-clearance ≥ 30 ml/min.
* INR < 2.
* Intrahepatic treatment can be accomplished
* The patients is approved by a multidisciplinary team

Exclusion Criteria:• Other current or prior malignant disease except adequately treated and cured carcinoma in situ of the cervix or squamous cell carcinoma of the skin.

* Cytotoxic or experimental treatment within a 14 days period before start of trial medication
* The patient is not allowed to participate in other clinical trials.
* Any clinical symptoms suggesting peripheral neuropathy grade 2
* Other severe medical conditions
* Severe cardial disease or AMI < 1 year
* Presence of diseases preventing oral therapy
* Patients with uncontrolled infection
* Pregnant or lactating women
* Women capable of childbearing not using a sufficient method of birth control
* Patients not able to understand the treatment or to collaborate
* Prior serious or unsuspected reaction after treatment with fluoropyrimidine
* Known prior hypersensitivity reactions to the agents
* Interstitial pneumonitis or pulmonary fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-02-02 (Actual); Primary Completion 2016-02-18 (Actual); Study Completion 2016-02-18 (Actual)

PRIMARY OUTCOMES:
PFS | 6 months after last patient included
  Time from treatment start to progression or death.

SECONDARY OUTCOMES:
Response rate. | 6 months after last patient included
Survival | 6 months after last patient included
Toxicity | 28 days after last treatment of last patient

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Bergenfeldt, Consultan, Principal Investigator — Department og Gastroenterology
Locations (1):
- Herlev Hospital, Herlev, Denmark